CLINICAL TRIAL: NCT05762497
Title: Pilot Feasibility Study of a Moldable Peristomal Adhesive for Pulmonary and Speech Rehabilitation After Total Laryngectomy
Brief Title: Pilot Feasibility Study of Peristomal Adhesives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Parrilla Claudio, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4650
Record Dates: First submitted 2023-02-17; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Laryngectomy; Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laryngectomized patients (Experimental)
  Interventions: Other: Moldable adhesive

INTERVENTIONS:
Other: Moldable adhesive — Patients were provided with the new adhesives and a short questionnaire on current ASV use. After a week, they were contacted by telephone to verify any doubts/problems. At the end of the two weeks, the patient was again administered a questionnaire to evaluate the new moldable adhesive (while using the ASV).

SUMMARY:
Loss of voice is one of the greater consequences of total laryngectomy. The voice prosthesis allows the patients to speak again in a very short time but forces them to use one hand when speaking. In order to reduce this discomfort and to allow "hands-free" speaking, an Automatic Speaking Valve (ASV) has been designed which is positioned on a peristomal adhesive.

Peristomal adhesives, however, tend to detach under the influence of mucus, cough, or phonatory pressure. Consequently, the current regular use of the automatic speaking valve in laryngectomees is very low. As a possible solution, Atos Medical AB has developed a moldable peristomal adhesive made of a thermoplastic elastomer, which becomes transparent and moldable when heated and facilitates precise contouring in situ. As the material cools, it loses its malleability but retains the integrity of the molded shape.

The expectation was that the moldable adhesive would provide a better individual fit and therefore longer fixation (especially when using the ASV).

To study the feasibility of this device, 10 total laryngectomized patients were asked to use the new moldable peristomal adhesive for two weeks in conjunction with their normal daily routine for adhesive application and removal, and speech rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Have undergone total laryngectomy
* Over the age of 18
* voice prosthesis user
* Experience in the use of adhesive and HMEs
* At least 3 months after total laryngectomy
* At least 6 months after the end of adjuvant radiotherapy
* Signature of the informed consent

Exclusion Criteria:

* Medical issues that prevent the use of HMEs and/or adhesives
* Recurrent or metastatic active disease
* Reduced mobility of the arms and/or hands
* Inability to understand the information and/or to provide informed consent
* Insufficient cognitive ability to handle HME or moldable adhesive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Investigation about product performance | 2 weeks
  Adhesive lifetime during hands-free speech use [hours]
Investigation about product performance | 2 weeks
  Use of hands-free speech [days/week]
Investigation about product performance | 2 weeks
  Duration of hands-free speech [hours/day]

SECONDARY OUTCOMES:
Parameters were expected to influence product performance and patient preference | 2 weeks
  Satisfaction (scored on a 5-point Likert scale)
Parameters were expected to influence product performance and patient preference | 2 weeks
  Adhesives fit (scored on a 5-point Likert scale)
Parameters were expected to influence product performance and patient preference | 2 weeks
  Adhesives usability (scored on a 5-point Likert scale),

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Parrilla, MD, PhD, Principal Investigator — Fondazione Policlinico Gemelli - IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli - IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No